CLINICAL TRIAL: NCT01265108
Title: Effects of Intravenous Iron Supplementation on Exercise Capacity During Sustained Alveolar Hypoxia in Healthy Humans.
Brief Title: Effects of Iron on Exercise Capacity During Hypoxia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: OHSRC-986
Record Dates: First submitted 2010-12-21; First posted 2010-12-22 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ferric Oxide, Saccharated; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous iron sucrose (Experimental): Infusion of 200 mg iron sucrose (Venofer) in 100 ml normal (0.9%) saline.
  Interventions: Drug: Iron sucrose.
- Intravenous normal saline (Placebo Comparator): Infusion of 100 ml normal (0.9%) saline.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Iron sucrose. — Volunteers will receive an intravenous infusion of 200 mg iron sucrose, before exposure to 8 hours of alveolar hypoxia. At the end of the exposure, pulmonary artery systolic pressure will be measured and volunteers will undertake an exercise test while breathing hypoxic gas.
  Other Names: Iron sucrose = Venofer
  Arms: Intravenous iron sucrose
Drug: Normal saline — Volunteers will receive an intravenous infusion of 100 ml normal saline, before exposure to 8 hours of alveolar hypoxia. At the end of the exposure, pulmonary artery systolic pressure will be measured and volunteers will undertake an exercise test while breathing hypoxic gas.
  Arms: Intravenous normal saline

SUMMARY:
During alveolar hypoxia, for example at high altitude or in patients with respiratory disease, there is evidence to suggest that hypoxia-induced pulmonary hypertension might limit exercise performance. Intravenous iron supplementation has recently been shown to reverse pulmonary hypertension in healthy humans at high altitude, and to prevent pulmonary hypertension in volunteers exposed to hypoxia at sea level. The investigators hypothesized that intravenous iron supplementation would enhance exercise capacity during alveolar hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Sea level natives with no recent exposure to high altitude
* Baseline iron indices within the normal range
* Detectable tricuspid regurgitation on echocardiography

Exclusion Criteria:

* Significant cardiorespiratory disease
* Known susceptibility to high altitude-related illness
* Taking medications or iron supplementation
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Maximal exercise capacity during hypoxia, assessed by maximal oxygen consumption. | After 8-h exposure to alveolar hypoxia.
  Volunteers will receive either intravenous iron or saline placebo, before exposure to 8 hours of alveolar hypoxia. They will then undergo an exercise test while breathing an hypoxic gas mixture. The primary outcome measure will be exercise capacity as determined by maximal oxygen consumption during this test. Volunteers will receive both interventions, via a crossover design. Due to uncertainty about the duration of action of iron at a cellular level, all volunteers will receive saline infusion on the first study day, and iron sucrose infusion on a second study day, at least one week later.

SECONDARY OUTCOMES:
Maximal exercise capacity, assessed by peak power output. | After 8-h exposure to alveolar hypoxia.
Pulmonary artery systolic pressure. | After 8-h exposure to alveolar hypoxia.
Blood levels of oxygen-regulated proteins. | After 8-h exposure to alveolar hypoxia

CONTACTS AND LOCATIONS:
Overall Officials: Nick P Talbot, DPhil MRCP, Principal Investigator — University of Oxford
Locations (1):
- Department of Physiology, Anatomy & Genetics, University of Oxford, Oxford, United Kingdom